CLINICAL TRIAL: NCT02426905
Title: Multicentre, Retrospective and Prospective Study to Assess Long-Term Outcomes of Chelator-Based Treatment With Trientine in Wilson Disease Patients Withdrawn From Therapy With d-Penicillamine
Brief Title: Study to Assess Long-Term Outcomes of Trientine in Wilson Disease Patients Withdrawn From Therapy With d-Penicillamine
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Univar BV (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UNV-TRI-002
Record Dates: First submitted 2014-09-18; First posted 2015-04-27 (Estimated); Last update posted 2017-08-23 (Actual); Status verified 2017-08

CONDITIONS: Wilson Disease
MeSH Terms: conditions — Hepatolenticular Degeneration | interventions — Trientine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Retrospective (No Intervention)
- Prospective (Other)
  Interventions: Drug: trientine dihydrochloride

INTERVENTIONS:
Drug: trientine dihydrochloride — A retrospective review of patients' medical records
  Arms: Prospective

SUMMARY:
A study to review Wilson disease patients who have previously been prescribed d- Penicillamine but were changed to trientine as treatment for their disease, and to follow them for a further 12 months.

DETAILED DESCRIPTION:
A retrospective study to review Wilson disease patients who have previously been prescribed d- Penicillamine but were changed to trientine as treatment for their disease, and to follow them prospectively for a further 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 1 year to 90 years of age.
* Physician established diagnosis of Wilson disease based on a Ferenci score > 3.
* Documented treatment with d-Penicillamine, withdrawal of treatment with d- Penicillamine, followed by treatment with trientine for at least 6 months at date of informed consent.
* Able/willing to provide written informed consent.
* For enrolment in the prospective part, enrolment in the retrospective part of the study is required.

Exclusion Criteria:

* Incomplete history of medication use for trientine from initial diagnosis to latest follow up.
* Unavailable outcome data for hepatic and neurological course of disease at assessment time points.
* Patients with acute liver failure and fulminant hepatic disease with fatal outcome.
* Hypersensitivity to trientine and severe anaemia.

Ages: 1 Year to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2016-01; Primary Completion 2018-05 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Clinical outcome specific to the retrospective part of the study | 48 months
  The clinical course of neurological and hepatic disease for each available time point after initiation of treatment (6, 12, 24, 36, and 48 months, and at the last available time point while taking second line trientine) will be scored (Investigator's score) based on neurological and hepatic status at the time of initiating trientine as: 1 = Unchanged 2 = Improved but not normal 3 = Improved to normal 4 = Asymptomatic over duration of therapy 5 = Worsened.
Clinical outcome specific to the prospective part of the study | 12 months
  The clinical course of neurological and hepatic disease will be scored (Investigator's score) based on the status at 6 and 12 months after Baseline as: 1 = Unchanged 2 = Improved but not normal 3 = Improved to normal 4 = Asymptomatic over duration of therapy 5 = Worsened A patient will be counted as a responder if they have a rating of ≤4 at the 12 month visit for both the neurological and hepatic Investigator's score. They will be counted as a non-responder if they have a rating = 5 for one or both scores at the 12 month visit or if they were discontinued from the study for any reason prior to the 12 month visit.

SECONDARY OUTCOMES:
Safety Endpoint Applicable to both the Retrospective and Prospective Parts of the Study | Up to 60 months
  All AEs related to trientine treatment, and AEs leading to discontinuation of trientine will be assessed at each available study time point.
Quality of Life Endpoints for the Prospective Part of the Study | 12 months
  The QoL questionnaires will be completed for each time point and data will be compared to baseline (prospective part) after 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Karl-Heinz Weiss, MD, Principal Investigator — Universitätsklinik Heidelberg
Locations (4):
- Universitätsklinik Heidelberg, Heidelberg, Germany
- "Aghia Sophia" Children's Hospital, Goudi, Greece
- San Paolo Hospital UOC, Milan, Italy
- Kings College Hospital, London, United Kingdom

REFERENCES:
- [Derived] Mohr I, Kruse C, Aliane V, Weiss KH. Prospective Study to Assess Long-Term Outcomes of Chelator-Based Treatment With Trientine Dihydrochloride in Patients With Wilson Disease. JGH Open. 2025 Mar 17;9(3):e70114. doi: 10.1002/jgh3.70114. eCollection 2025 Mar. PMID 40104015
- [Derived] Weiss KH, Kruse C, Manolaki N, Zuin M, Ferenci P, van Scheppingen D, Wijnberg L, de Koning CE, Dhawan A. Multicentre, retrospective study to assess long-term outcomes of chelator based treatment with trientine in Wilson disease patients withdrawn from therapy with d -penicillamine. Eur J Gastroenterol Hepatol. 2022 Sep 1;34(9):940-947. doi: 10.1097/MEG.0000000000002387. Epub 2022 Apr 29. PMID 35482910